CLINICAL TRIAL: NCT02147964
Title: Mechanisms of Hormonal Control of Spermatogenesis in Man
Brief Title: ITT-5 Mechanisms of Spermatogenesis in Man
Acronym: ITT-5
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding was obtained for this study.
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, William Bremner, Professor of Medicine, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001449
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Gonadotropin Deficiency
Keywords: intratesticular androgens; testosterone; dutasteride; gonadotropin suppression; male contraception; spermatogenesis
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; Gels; Coal Tar; acyline; Dutasteride; Ketoconazole; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Acyline; T Gel; placebo dutasteride, placebo ketoconazole (Experimental): All men will receive Acyline 300 ug/kg subcutaneous (SQ) injections every 2-weeks + Testosterone 1% Gel 5g daily and then randomly assigned.
  Group 1: placebo oral ketoconazole + placebo oral dutasteride for 4 months
  Interventions: Drug: Testosterone 1% Gel; Drug: Acyline; Drug: placebo dutasteride; Drug: placebo ketoconazole
- Acyline; T gel; Ketoconazole; placebo (Experimental): All men will receive Acyline 300 ug/kg SQ injections every 2-weeks + Testosterone 1% Gel 5g daily and then randomly assigned.
  Group 2: oral ketoconazole 400 mg + placebo oral dutasteride for 4 months
  Interventions: Drug: Testosterone 1% Gel; Drug: Acyline; Drug: Ketoconazole; Drug: placebo dutasteride
- Acyline; Tgel; Ketoconazole; Dutasteride (Experimental): All men will receive Acyline 300 ug/kg SQ injections every 2-weeks + Testosterone 1% Gel 5g daily and then randomly assigned.
  Group 3: Ketoconazole 400mg orally daily + Dutasteride 2.5 mg orally on day 1, followed by 0.5mg daily for 4 months
  Interventions: Drug: Testosterone 1% Gel; Drug: Acyline; Drug: Dutasteride; Drug: Ketoconazole
- Acyline; Tgel; HCG (Experimental): All men will receive Acyline 300 ug/kg SQ injections every 2-weeks + Testosterone 1% Gel 5g daily and then randomly assigned.
  Group 4: Human Chorionic gonadotropin (HCG) 60 IU injection every other day for 4 months.
  Interventions: Drug: Testosterone 1% Gel; Drug: Acyline; Drug: HCG

INTERVENTIONS:
Drug: Testosterone 1% Gel — Testosterone 1% gel 5g daily for 4 months [all subjects]
  Other Names: T gel; Testosterone gel; AndroGel
Drug: Acyline — Acyline 300 ug/kg SQ injections every 2-weeks for 4 months [all subjects]
Drug: Dutasteride — Dutasteride 2.5 mg (day 1) followed by 0.5 mg daily for 4 months
  Other Names: Avodart
  Arms: Acyline; Tgel; Ketoconazole; Dutasteride
Drug: Ketoconazole — ketoconazole 400 mg PO daily for 4 months
  Arms: Acyline; T gel; Ketoconazole; placebo; Acyline; Tgel; Ketoconazole; Dutasteride
Drug: HCG — HCG 60 IU injection Subcutaneously, every other day for 4 months
  Other Names: Human chorionic gonadotropin (HCG)
  Arms: Acyline; Tgel; HCG
Drug: placebo dutasteride — placebo oral dutasteride PO daily for 4 months
  Arms: Acyline; T Gel; placebo dutasteride, placebo ketoconazole; Acyline; T gel; Ketoconazole; placebo
Drug: placebo ketoconazole — placebo ketoconazole daily for 4 months
  Arms: Acyline; T Gel; placebo dutasteride, placebo ketoconazole

SUMMARY:
The purpose of this investigational drug study is to determine how much male hormone, testosterone, is needed to maintain sperm production in the testis.

DETAILED DESCRIPTION:
This is a nine-month research study examining the effects on androgen treatment on sperm production in healthy men. There are three phase to the study, a 2-month screening phase, 4-month treatment and 3-month follow-up. In this study, the investigators aim to define a quantitative relationship between intra-testicular testosterone (IT-T) and spermatogenesis in man. Hormone levels will be measured in a small amount of testicular fluid at the beginning and end of treatment and sperm concentration will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18-55
* In general good health based on normal screening evaluation
* Normal serum testosterone, lutenizing hormone (LH) and follicle stimulating hormone (FSH)
* Prostate Specific Antigen (PSA) < 3.0
* Agrees not to donate blood or participate in another research study during the study
* Informed consent
* Must be willing to use a reliable form of contraception during the study

Exclusion Criteria:

* Participation in a long-term male contraceptive study within the past three months
* History of testosterone or anabolic steroid abuse in the past
* History of or current skin disorder that will interfere with testosterone gel
* Poor general health or significantly abnormal screening blood results
* History of or current testicular or prostate disease
* History of a bleeding disorder or need for anticoagulation
* History of untreated sleep apnea and/or major psychiatric problems
* BMI > 32
* History of or current liver disease
* Chronic pain syndrome
* Current use of terfenidine, astemizole, cisapride, budesonide, felodipine, fluticasone, lovastatin, midazolam, sildenafil, or vardenafil
* Use of glucocorticoids or underlying adrenal insufficiency
* Active drug or alcohol abuse within the past year

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sperm concentration | 16 weeks
  Difference in sperm concentration at week 16 between 4 treatment groups

SECONDARY OUTCOMES:
IT steroid concentration | 16 weeks
  It steroid concentration at week 16 between the 4 treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Mara Roth, MD, Principal Investigator — University of Washington; William J Bremner, MD, PhD, Study Director — University of Washington
Locations (1):
- University of Washington Medical Center (Health Sciences), Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Contraceptive efficacy of testosterone-induced azoospermia in normal men. World Health Organization Task Force on methods for the regulation of male fertility. Lancet. 1990 Oct 20;336(8721):955-9. PMID 1977002
- [Background] Wu FC, Farley TM, Peregoudov A, Waites GM. Effects of testosterone enanthate in normal men: experience from a multicenter contraceptive efficacy study. World Health Organization Task Force on Methods for the Regulation of Male Fertility. Fertil Steril. 1996 Mar;65(3):626-36. PMID 8774299
- [Background] Anawalt BD, Bebb RA, Bremner WJ, Matsumoto AM. A lower dosage levonorgestrel and testosterone combination effectively suppresses spermatogenesis and circulating gonadotropin levels with fewer metabolic effects than higher dosage combinations. J Androl. 1999 May-Jun;20(3):407-14. PMID 10386821
- [Background] Zirkin BR, Santulli R, Awoniyi CA, Ewing LL. Maintenance of advanced spermatogenic cells in the adult rat testis: quantitative relationship to testosterone concentration within the testis. Endocrinology. 1989 Jun;124(6):3043-9. doi: 10.1210/endo-124-6-3043. PMID 2498065
- [Background] Roth MY, Lin K, Amory JK, Matsumoto AM, Anawalt BD, Snyder CN, Kalhorn TF, Bremner WJ, Page ST. Serum LH correlates highly with intratesticular steroid levels in normal men. J Androl. 2010 Mar-Apr;31(2):138-45. doi: 10.2164/jandrol.109.008391. Epub 2009 Sep 24. PMID 19779211
- [Background] Roth MY, Page ST, Lin K, Anawalt BD, Matsumoto AM, Snyder CN, Marck BT, Bremner WJ, Amory JK. Dose-dependent increase in intratesticular testosterone by very low-dose human chorionic gonadotropin in normal men with experimental gonadotropin deficiency. J Clin Endocrinol Metab. 2010 Aug;95(8):3806-13. doi: 10.1210/jc.2010-0360. Epub 2010 May 19. PMID 20484472
- [Background] Trachtenberg J, Zadra J. Steroid synthesis inhibition by ketoconazole: sites of action. Clin Invest Med. 1988 Feb;11(1):1-5. PMID 2966691
- [Background] Nashan D, Knuth UA, Weidinger G, Nieschlag E. The antimycotic drug terbinafine in contrast to ketoconazole lacks acute effects on the pituitary-testicular function of healthy men: a placebo-controlled double-blind trial. Acta Endocrinol (Copenh). 1989 May;120(5):677-81. doi: 10.1530/acta.0.1200677. PMID 2499150
- [Background] Pont A, Graybill JR, Craven PC, Galgiani JN, Dismukes WE, Reitz RE, Stevens DA. High-dose ketoconazole therapy and adrenal and testicular function in humans. Arch Intern Med. 1984 Nov;144(11):2150-3. PMID 6093722
- [Background] Van Tyle JH. Ketoconazole. Mechanism of action, spectrum of activity, pharmacokinetics, drug interactions, adverse reactions and therapeutic use. Pharmacotherapy. 1984 Nov-Dec;4(6):343-73. doi: 10.1002/j.1875-9114.1984.tb03398.x. PMID 6151171
- [Background] Roth MY, Nya-Ngatchou JJ, Lin K, Page ST, Anawalt BD, Matsumoto AM, Marck BT, Bremner WJ, Amory JK. Androgen synthesis in the gonadotropin-suppressed human testes can be markedly suppressed by ketoconazole. J Clin Endocrinol Metab. 2013 Mar;98(3):1198-206. doi: 10.1210/jc.2012-3527. Epub 2013 Jan 24. PMID 23348398
- [Background] Coviello AD, Matsumoto AM, Bremner WJ, Herbst KL, Amory JK, Anawalt BD, Sutton PR, Wright WW, Brown TR, Yan X, Zirkin BR, Jarow JP. Low-dose human chorionic gonadotropin maintains intratesticular testosterone in normal men with testosterone-induced gonadotropin suppression. J Clin Endocrinol Metab. 2005 May;90(5):2595-602. doi: 10.1210/jc.2004-0802. Epub 2005 Feb 15. PMID 15713727